CLINICAL TRIAL: NCT04954924
Title: Acute and Long Term Effect of Kinesio Tape on Motor Function, Proprioception and Balance in Subjects With ACL Rupture
Brief Title: Effect of Kinesio Tape on Motor Function in Subjects With ACL Rupture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LithuananianSportsU-6
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: ACL Rupture; Rehabilitation
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group - standardized physiotherapy program (No Intervention): The standardized physiotherapy program was designed on the basis of S. van Grinsven et al.'s (2010) rehabilitation protocol - was applied 4 weeks, 3 times per week, the duration of the procedure was 60 minutes.
- Experimental group - standardized physiotherapy program and Kinesio tape (Experimental): The standardized physiotherapy program was designed on the basis of S. van Grinsven et al.'s (2010) rehabilitation protocol - was applied 4 weeks, 3 times per week, the duration of the procedure was 60 minutes. The Kinesio tape (KT) technique was chosen on the basis of K. Kase et al.'s (2003) recommendations. KT (Japan) was applied to the injured leg using muscular and functional-corrective techniques on the quadriceps femoris and the hamstring muscle. There were 6 KT procedures per participant in the experimental group. The CON group received KT only during the baseline and final assessment to assess short-term effect of KT.
  Interventions: Other: standardized physiotherapy program and Kinesio tape

INTERVENTIONS:
Other: standardized physiotherapy program and Kinesio tape
  Arms: Experimental group - standardized physiotherapy program and Kinesio tape

SUMMARY:
Thirty-two participants with ACL rupture were included in the study. All participants were divided in two groups - control and experimental. In the experimental group (n=16) participants received 4 weeks standardized physiotherapy and Kinesio tape, in the control group - standardized physiotherapy.

Experimental measurements: Anthropometric measurements, pain intensity, static and dynamic balance, proprioception, knee flexion and extension muscle torque, level of activity

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 35-year-old men;
2. a normal contralateral knee,
3. not a longer period than 3 months after ACL rupture.

Exclusion Criteria:

Participants were excluded if either knee had previously been injured or had undergone surgery, if they had concurrent osteoarthritis, if they had injured the posterior cruciate ligament, lateral collateral ligament, or posterolateral complex of the knee, or if they had a grade III tear of the medial collateral ligament.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2015-01-15 (Actual); Study Completion 2015-01-15 (Actual)

PRIMARY OUTCOMES:
Static and dynamic balance | 4 weeks
  Static and dynamic balance were measured by posturography method with a single piezoelectric force plate (KISTLER, Switzerland, Slimline System 9286) was used to measure postural sway activity.
Muscle torque | 4 weeks
  The isometric and concentric torque of the knee extensor and flexor muscles of the non-injured and injured legs was measured using an isokinetic dynamometer (System 3; Biodex Medical Systems, Shirley, New York).
Joint position sense test | 4 weeks
  Joint position sense test was used to measure proprioceptive accuracy. Joint position sense for both legs was assessed for all subjects using the Biodex System Isokinetic Dynamometer 3 (Biodex Medical System Inc., Shirley, NY, USA).Subjects actively extended the knee from the resting position (90°flexion) to one of two test positions: 80° or 40° flexion at 0,5°/s velocity. Subjects were instructed to actively reproduce this criterion angle and to stop knee motion, via a thumb switch. No feedback was provided.

SECONDARY OUTCOMES:
The Lysholm scale | 4 weeks
  The Lysholm scale does measure the domains of symptoms and complaints and does measure functioning in daily activities
The Tegner scale | 4 weeks
  The Tegner scale measure the subjective functional activity
VAS scale | 4 weeks
  The severity of pain was determined based on a numerical pain scale in which 0 symbolizes 'no pain' and 10 symbolizes 'maximum pain'

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiele D, Solianik R. Four-Week Application of Kinesiotaping Improves Proprioception, Strength, and Balance in Individuals With Complete Anterior Cruciate Ligament Rupture. J Strength Cond Res. 2023 Jan 1;37(1):213-219. doi: 10.1519/JSC.0000000000004245. Epub 2022 Apr 13. PMID 35438677